CLINICAL TRIAL: NCT04579237
Title: Development and Evaluation of Techniques for Computer Aided Detection and Diagnosis From Existing Radiologic Images
Status: Active, not recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000037; 000037-CC
Record Dates: First submitted 2020-10-07; First posted 2020-10-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09-26

CONDITIONS: Radiology Information Systems
Keywords: Opportunistic screening; Artificial Intelligence; Automated Detection; Epidural Masses; Lymphadenopathy; Natural History
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/All Subjects: Data will be derived from primary studies on all subjects.

SUMMARY:
Background:

Radiologic images are getting more complex. They are also being used more often. Medical personnel are overwhelmed with data. Computer Aided Detection (CAD) and diagnosis may be able to improve medical care. Researchers want to create and test ways to use CAD. To do this, they want to use data from the Clinical Center s Department of Diagnostic Radiology.

Objective:

To create algorithms and software that accurately detect and characterize lesions, model anatomy, and monitor diseases on radiologic studies.

Eligibility:

People of all ages who have radiologic exams stored in the clinical PACS (picture archiving system) of the Clinical Center since July 6, 1953 with no end date. People with target lesions of any kind will be included.

Design:

This study will use existing data. Participants will include males and females of all ages. They will be chosen by keyword search on NIH databases.

The data that is used may include CT, MRI, ultrasound, and other images. It may include a participant s name, date of birth, and date of exam. It may include the name of the doctor, radiologist, and hospital. Data such as age, gender, race, disease, and treatment may be used. Other data from charts or studies may be used.

Imaging data of all organs of the body will be studied.

Data will be kept in computers and servers. The equipment will be password protected. Printouts will be stored in locked rooms.

This study will last 10 years.

DETAILED DESCRIPTION:
Study Description:

This study uses artificial intelligence techniques to improve radiology diagnosis.

Objective:

Development of Computer Aided Detection techniques to improve radiology imaging.

Study Population:

Up to 1,000,000 NIH Clinical Center patients.

Description of Sites/Facilities conducting research:

NIH Clinical Center

Study Duration:

10 years

ELIGIBILITY:
* INCLUSION CRITERIA:
* All radiologic exams available in the clinical PACS (picture archiving system) of the Clinical Center taken from July, 6, 1953 with no end date.
* Males and Females of all ages.
* Patients with target lesions of any kind will be included
* Patients without the target lesion will be included to determine the specificity of the computer aided detection or diagnosis algorithm

EXCLUSION CRITERIA:

None

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Special classes of subjects, such as pregnant women, children, cognitively impaired individuals, or others likely to be vulnerable will be included since the data has already been obtained under an IRB-approved protocol and there are no anticipated additional risks from this research
Sampling Method: Probability Sample
Enrollment: 144625 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Development of Computer Aided Detection techniques to improve radiology imaging | End of study
  Development of Computer Aided Detection techniques to improve radiology imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Summers, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000037-CC.html